CLINICAL TRIAL: NCT06830473
Title: KTRSensor Scotland Study: Investigating the Role of Biomarkers in Kidney Transplant Outcomes
Brief Title: KTRSensor Scotland Study: An Observational Study Into Predictors and Diagnosis of Kidney Transplant Rejection
Acronym: KTRSensors
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC24216
Record Dates: First submitted 2025-02-05; First posted 2025-02-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Kidney Transplant; Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Routine collection of midstream urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational study capturing real world transplant patients in the post-operative setting aiming to further determine the utility of biomarkers to improve outcomes.

DETAILED DESCRIPTION:
A prospective longitudinal observational study capturing patients receiving kidney transplants in Scotland. The primary objective is to assess whether there are clinical biomarkers present in the urine that determine the outcome of kidney transplants and predict early graft rejection.

ELIGIBILITY:
Any patient within a Scottish Transplant centre who has undergone renal transplant (+/- pancreas/islet) and is due to attend routine follow-up appointments at the index centre.

Exclusion criteria:

* no previous kidney transplant
* patient attending follow-up at a peripheral site
* unable to provide urine samples across the study duration

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population sampled from those who have recently undergone renal transplant in a Scottish transplant centre
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2028-05-13 (Estimated); Study Completion 2028-05-13 (Estimated)

PRIMARY OUTCOMES:
Number of participants that experience acute transplant rejection | 12 months
  Defined by gold standard core biopsy, reported using the Banff histology grading.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Vendrell, PhD, Study Chair — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - Royal Infirmary of Edinburgh, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow

IPD SHARING:
Plan to Share IPD: No